CLINICAL TRIAL: NCT03841422
Title: Evaluation of Video-assisted Instructions of Nasal Self-packing in Patients with Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Evaluation of Video-assisted Instructions of Nasal Self-packing in Patients with HHT
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Freya Droege, Principle Investigator, University Hospital, Essen
Other Study IDs: Nasal self-packing in HHT
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Haemorrhagic Telangiectasia
Keywords: hereditary hemorrhagic telangiectasia; video-assisted teaching; nasal self-packing
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: video-assisted nasal self-packing — video-assisted nasal self-packing

SUMMARY:
Inserting nasal self-packings is a secure method leaving patients more self-confident. We provide a video on https://www.youtube.com/watch?v=LaioLYfSJ-E demonstrating how to use nasal self-packings.

DETAILED DESCRIPTION:
Inserting nasal self-packings is a secure method leaving patients more self-confident. In HHT centers, patients often learn how to use them, but these centers are rare. Providing a video on https://www.youtube.com/watch?v=LaioLYfSJ-E demonstrating how to use nasal self-packings may also help patients without access to HHT centers.

ELIGIBILITY:
Inclusion Criteria:

* age above 17 years old

Exclusion Criteria:

* patients younger than 18 years old
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hereditary hemorrhagic telangiectasia who often suffer from recurrent nosebleeds
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of video-assisted teaching | 1 year
  Evaluation of video-assisted teaching using a questionnaire. Data about using new media (Do you use a smartphone/ tablet (yes/no)? Do you use the internet (e.g. youtube, facebook, instagram...)?) Moreover, patients feeling loosing control (before and after using pneumatic nasal self-packing: how often do have the feeling of losing control (scale form 1 to 5, 1 = very often, 5 = never) and safety (after learning the nasal self-packing with pneumatic tamponades do you feel safe? (scale 1 to 5, 1 = not very safe, 5 = safe) is analyzed. Additional data about number of blood transfusions, hospitalty and doctoral consulation rates (regarding recurrent nosebleeds in the last 12 months: How many bloodtranfusions did you get (because of nosebleeds/ gastrointestinal bleedings/ both)? How often did you see a doctor or needed to be treated in hospital?) is documented.

SECONDARY OUTCOMES:
Analyzing duration of consultation | 1 year
  the duration of the consultation and seeing the video is documented and compared to the Duration of consultations in patients with HHT before having uploaded the video

CONTACTS AND LOCATIONS:
Overall Officials: Freya Droege, Dr. med., Principal Investigator — University Hospital, Essen; Freya Droege, Dr. med., Study Chair — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, Nordrhein Westphalen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shovlin CL, Guttmacher AE, Buscarini E, Faughnan ME, Hyland RH, Westermann CJ, Kjeldsen AD, Plauchu H. Diagnostic criteria for hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber syndrome). Am J Med Genet. 2000 Mar 6;91(1):66-7. doi: 10.1002/(sici)1096-8628(20000306)91:13.0.co;2-p. PMID 10751092
- [Background] Droege F, Lueb C, Thangavelu K, Stuck BA, Lang S, Geisthoff U. Nasal self-packing for epistaxis in Hereditary Hemorrhagic Telangiectasia increases quality of life. Rhinology. 2019 Jun 1;57(3):231-239. doi: 10.4193/Rhin18.141. PMID 30739126
- [Background] Faughnan ME, Palda VA, Garcia-Tsao G, Geisthoff UW, McDonald J, Proctor DD, Spears J, Brown DH, Buscarini E, Chesnutt MS, Cottin V, Ganguly A, Gossage JR, Guttmacher AE, Hyland RH, Kennedy SJ, Korzenik J, Mager JJ, Ozanne AP, Piccirillo JF, Picus D, Plauchu H, Porteous ME, Pyeritz RE, Ross DA, Sabba C, Swanson K, Terry P, Wallace MC, Westermann CJ, White RI, Young LH, Zarrabeitia R; HHT Foundation International - Guidelines Working Group. International guidelines for the diagnosis and management of hereditary haemorrhagic telangiectasia. J Med Genet. 2011 Feb;48(2):73-87. doi: 10.1136/jmg.2009.069013. Epub 2009 Jun 23. PMID 19553198
- See also: video about using nasal self-packings — https://www.youtube.com/watch?v=LaioLYfSJ-E